CLINICAL TRIAL: NCT02481544
Title: The Effects of Journaling on Health-Related Mood and Clinical Outcomes in Post-MI Patients
Acronym: GRAT2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul J. Mills, Professor IR, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R21AT008033-01A1 (NIH)
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Myocardial Infarction; Psychosocial Factors
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gratitude Journaling Plus Standard of Care (Experimental): The most often used gratitude intervention consists of journaling, writing lists of things for which the individual is grateful. This technique was first employed and found to be effectual for enhancing wellbeing by Emmons and McCullough and has been suggested to be as effective as methods frequently used in clinical therapy. We are proposing an 8-week intervention in which the participant records 3-5 things for which they are grateful most days of the week. A longer intervention was chosen because Emmons and McCullough (2003) suggest that healthy behavior changes only occurred in a prolonged multi-week intervention. To ensure some conformity in the intervention, instructions that will be used will be similar to Emmons and McCullough (2003): "There are many things in our lives, both large and small, that we might be grateful about. Think back over your day (week) and write down on the lines below up to five things in your life that you are grateful or thankful for."
  Interventions: Behavioral: Gratitude Journaling Plus SOC
- Memorable Events Journaling Plus Standard of Care (Sham Comparator): In the sham control condition, individuals will record "memorable events" with methods identical to the gratitude journaling condition: Patients will be asked to record 3-5 memorable events in a given day, on most days of the week. Patients will be contacted once per week to remind them to continue with the memorable events journal. Patients will be given 2 journals during their first testing session (one journal is for the first four weeks and the second is for the second four weeks of journaling). Patients will be contacted once per week to remind them to continue with gratitude journal writing. Patients will be instructed to record the date of each journal entry next to each new day of journaling Patients will be provided with materials to return their first journal by mail and will and return their second journal at the T2 laboratory testing session.
  Interventions: Behavioral: Memorable Events Journaling Plus SOC
- Standard of Care (No Intervention): SOC consists of medical care that is included in post-MI treatment, such as physician visits and medication adjustments and cardiac rehabilitation. These patients will not have any active intervention, but will undergo the same testing routine as the gratitude intervention group. These patients will be given the opportunity to participate in the gratitude journaling intervention after they have completed the study. Patient records will be evaluated at each timepoint for changes in medications and medical treatment.

INTERVENTIONS:
Behavioral: Gratitude Journaling Plus SOC
  Arms: Gratitude Journaling Plus Standard of Care
Behavioral: Memorable Events Journaling Plus SOC
  Arms: Memorable Events Journaling Plus Standard of Care

SUMMARY:
Psychosocial factors, including positive affect, finding meaning in the event, and managing emotional distress, influence prognosis following a heart attack or myocardial infarction (MI). Gratitude, typically defined as a feeling or attitude in acknowledgment of a benefit that one has received or will receive, is associated with higher levels of well-being, and people who are more grateful experience less stress, are less depressed, have higher levels of control over their environment, and more positive ways of coping. The present project will examine the potential benefits of a gratitude intervention (i.e., 8 weeks of gratitude journaling) to increase positive health behaviors, psychological health, and physical functioning in post-MI patients as compared to journaling about memorable events as well as care as usual alone. The investigators will study psychological and physical functioning at baseline, following 8 weeks of gratitude journaling or care as usual, and at 4-month follow-up.

ELIGIBILITY:
Inclusion criteria:

1. Suffered an MI (ST Elevation MI (STEMI) or Non-ST Elevation MI (NSTEMI) with creatine kinase MB fraction elevation 3 times the upper limits of normal and with ischemic ECG changes within 12 months of baseline testing;
2. An EF less than 50% on echocardiogram;
3. Clinically stable defined as, no active arrhythmia, no residual ischemia;
4. Able to perform light to moderate exercise;
5. Able to give informed consent in English;
6. Medical clearance by their cardiologist;
7. > 35 years of age.

Exclusion criteria:

1. Unstable angina;
2. Severe valvular disease;
3. Oxygen-dependent COPD;
4. Recent stroke or significant cerebral neurologic impairment;
5. Suicidality with intent or plan;
6. Current cancer;
7. Currently taking mood stabilizers, benzodiazepines or antipsychotics;
8. Medications (e.g., systemic steroids) and conditions affecting immune status (e.g., rheumatoid arthritis, hepatitis C, HIV) (Anti-depressant medication is allowed);
9. Currently enrolled in another clinical trial.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by Recruitment rates will be recorded and new recruitment strategies will be formulated to overcome barriers presented by decliners for a future study. | 2 years
Treatment Expectancy & Satisfaction assessed by Treatment expectancy and satisfaction - 6 item credibility/ expectancy questionnaire (CEQ) will be utilized | 2 years
Retention assessed by Retention (% of drop-outs) will be recorded, and exit interviews will be administered to determine reasons for drop-out. | 2 years
Adherence assessed by Adherence to intervention will be derived from gratitude journals. | 2 years

SECONDARY OUTCOMES:
Gratitude | 2 years
  There are three scales that have been developed to measure gratitude, the Gratitude Questionnaire (GQ-6) (McCullough et al., 2002), Appreciation Scale (Adler & Fagley, 2005), and Gratitude, Appreciation, and Resentment Test (GRAT). Each scale came from a different concept of gratitude, and in concert they provide a broad definition of gratitude. According to Wood, Maltby, Stewart and Joseph (2008) the three scales comprise 12 sub-scales which measure eight different components of gratitude: (1) grateful affect, (2) appreciation of other people, (3) a focus on what the person has, (4) feelings of awe when encountering beauty, (4) behaviors to express gratitude, (5) focusing on the positive in the present moment, (6) appreciation rising from understanding life is short, (7) a focus on the positive in the present moment, and (8) positive social comparisons.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Peterson CT, Lucas J, John-Williams LS, Thompson JW, Moseley MA, Patel S, Peterson SN, Porter V, Schadt EE, Mills PJ, Tanzi RE, Doraiswamy PM, Chopra D. Identification of Altered Metabolomic Profiles Following a Panchakarma-based Ayurvedic Intervention in Healthy Subjects: The Self-Directed Biological Transformation Initiative (SBTI). Sci Rep. 2016 Sep 9;6:32609. doi: 10.1038/srep32609. PMID 27611967